CLINICAL TRIAL: NCT05956600
Title: An Open-Label, Single-Arm Clinical Trial Evaluating the Safety and Efficacy of Amisulpride in Treating Patients With Schizophrenia and Schizoaffective Disorder Who Have Treatment-Resistant Positive Symptoms
Acronym: AmisulprideTRS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Action of PI. Loss of sponsor
Sponsor: University of California, Los Angeles (Other)
Collaborators: PoloMar Health LLC (Industry)
Responsible Party: Principal Investigator, Stephen R. Marder, Professor of Psychiatry, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMI 1
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Schizophrenia, Treatment-Resistant
Keywords: Schizophrenia; Schizoaffective Disorder; Amisulpride
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant; Schizophrenia; Psychotic Disorders | interventions — Amisulpride

STUDY DESIGN:
Intervention Model Description: Single-Arm Administration of Amisulpride
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amisulpride (Other): Amisulpride administered orally. Dose range 50 to 1200 mg daily
  Interventions: Drug: Amisulpride 50 MG

INTERVENTIONS:
Drug: Amisulpride 50 MG — Amisulpride 50 mg titrated to dose range of 50 to 1200 mg

SUMMARY:
The objectives of this study are to evaluate the safety and efficacy of Amisulpride as an add-on therapy or alternative monotherapy in treating patients with schizophrenia or schizoaffective disorder who have treatment-resistant positive symptoms and who are not eligible for treatment with clozapine due to intolerance, failure from a prior clozapine trial, or unwillingness to be treated with clozapine.

DETAILED DESCRIPTION:
Prior to enrollment, eligible patients and their treating psychiatrist will decide whether the goal is to evaluate amisulpride as an antipsychotic that is added to the current medication or as an alternative monotherapy. All study participants will receive amisulpride in oral form.

For monotherapy patients, after primary and secondary endpoints are recorded, the study psychiatrist will begin a gradual cross-taper of the patient's current antipsychotic medication to amisulpride. The goal will be to have the patient on monotherapy by the one-month rating. The dose of amisulpride will vary depending on whether amisulpride will be used as an add-on therapy or monotherapy. The starting dose of amisulpride will be 50 mg/day and will be increased in 50 mg increments every 2-3 days until the optimal dose is reached, as determined by the treating psychiatrist, with a maximum dose of 1,200 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed and dated written informed consent. 2. Age 18-65 years 3. Male or female*. 4. *For participants assigned female sex at birth: A participant is eligible to participate if not pregnant, and one of the following conditions applies: (1) Is not able to become pregnant; (2) is a person able to be pregnant (PABP) and using a contraceptive method that is highly effective, with a failure rate of <1%.

  5. Diagnosis of schizophrenia or schizoaffective disorder according to DSM-V criteria 6. Treatment-resistant positive symptoms defined by subjects receiving an antipsychotic but continuing to score 4 or greater one of the following Positive and Negative Syndrome Scale (PANSS) items: P1 (delusions), P3 (hallucinations), P6 (suspiciousness or persecution), or G9 (unusual thought content).

  7. Subjects receiving clozapine will also be included if there is a concern that the side effect burden from clozapine has led the clinician and the patient to consider changing to another medication.

  8. English-speaking. 9. Subjects only partially responsive to other antipsychotics will also be included.

  10. Non-suicidal self-injurious behavior may be included if approved by the study clinician.

  11. Able to provide informed consent.

Exclusion Criteria:

1. Diagnosis of any other psychiatric disorder.
2. History of intolerance or allergy to amisulpride.
3. Known history of severe cardiac arrhythmia or prolonged QT interval.
4. Concomitant use of medications that may interact with amisulpride or prolong QT interval (see section 4.3, "Concomitant Therapy").
5. Lactating patients, patients with prolactin-dependent tumors, and patients with breast cancer will be excluded.
6. Patients with laboratory- and/or imaging-confirmed pheochromocytoma will be excluded.
7. Columbia-Suicide Severity Rating Scale:

   * Suicidal ideation score of 4 or greater within the last month of the assessment at a frequency of once a week or more.
   * Suicidal ideation score of 5 within the last 6 months of the assessment.
   * Any suicidal behavior, including suicide attempts or preparatory acts, within the last 6 months of the assessment.
8. Current moderate or severe alcohol and substance use disorders, which could pose a safety concern or interfere with the therapeutic process.
9. Existing relevant physical health problems: such as cardiovascular disease, previous problems with prolactin, impaired liver/renal function or epilepsy.
10. Any medical condition that the PI determines could jeopardize the safety of the study subject or compromise the integrity of the data.
11. Planning to start a new drug, diet, or behavioral intervention during the study.
12. A previous trial of amisulpride.
13. Unable to perform or cooperate with study requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Symptom Scale | Baseline to 12 months
  Change in Total Score

IPD SHARING:
Plan to Share IPD: Undecided